CLINICAL TRIAL: NCT00005465
Title: Genetic Mapping of Atherogenic Lipoprotein Phenotypes
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4909; R01HL046880 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2001-05

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases

SUMMARY:
To map the major gene influencing low-density lipoprotein subclass phenotypes, denoted atherogenic lipoprotein (ALP) phenotypes, with a long term goal of cloning the ALP gene and understanding its role in genetic susceptibility to atherosclerosis.

DETAILED DESCRIPTION:
BACKGROUND:

ALP phenotype B (ALP-B), characterized by a predominance of small, dense LDL particles as determined by gradient gel electrophoresis, has been associated with increased risk of myocardial infarction and a constellation of atherogenic lipid and apolipoprotein (apo) changes. Based on complex segregation analysis, ALP-B appeared to be influenced by a single major genetic locus with a dominant mode of inheritance and a common allele frequency. This project was designed to identify a new gene involved in susceptibility to coronary heart disease.

DESIGN NARRATIVE:

The investigators identified, collected and constructed a repository of immortalized cell lines and lipid and apo measurements from members of families informative for ALP. They tested genes implicated in lipoprotein metabolism as possible candidate ALP genes and used highly informative DNA probes to search the genome for linkage to the ALP gene. They also refined the model for the inheritance of ALP phenotypes and tested for genetic-environmental interactions. Forty informative families were recruited for the repository. The families were identified through two sources of probands: former participants in a cholesterol-lowering diet study and patients seen at the lipid clinics at the University of Washington. Each participating family member completed a medical history questionnaire and provided a blood sample for ALP phenotype determination, for DNA studies, and for lipid and apo measurements. Linkage studies and LOD score analyses began with a candidate gene approach, and continued by using DNA probes that revealed restriction fragment length polymorphisms (RFLPs) to search the genome for linkage to the ALP gene. When a linkage was found, ALP genotype information was used to refine the statistical model describing the inheritance of ALP phenotypes, and to evaluate genetic-environmental interactions involving lipid and apo levels and environmental and behavioral factors.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-08; Study Completion 1996-07

REFERENCES:
- [Background] Austin MA, Talmud PJ, Luong LA, Haddad L, Day IN, Newman B, Edwards KL, Krauss RM, Humphries SE. Candidate-gene studies of the atherogenic lipoprotein phenotype: a sib-pair linkage analysis of DZ women twins. Am J Hum Genet. 1998 Feb;62(2):406-19. doi: 10.1086/301712. PMID 9463319
- [Background] Austin MA. Genetic epidemiology of dyslipidaemia and atherosclerosis. Ann Med. 1996 Oct;28(5):459-63. doi: 10.3109/07853899608999108. PMID 8949979
- [Background] Austin MA, Edwards KL. Small, dense low density lipoproteins, the insulin resistance syndrome and noninsulin-dependent diabetes. Curr Opin Lipidol. 1996 Jun;7(3):167-71. doi: 10.1097/00041433-199606000-00010. PMID 8818515
- [Background] Austin MA, Selby JV. LDL subclass phenotypes and the risk factors of the insulin resistance syndrome. Int J Obes Relat Metab Disord. 1995 May;19 Suppl 1:S22-6. PMID 7550534
- [Background] Austin MA, Hokanson JE, Brunzell JD. Characterization of low-density lipoprotein subclasses: methodologic approaches and clinical relevance. Curr Opin Lipidol. 1994 Dec;5(6):395-403. doi: 10.1097/00041433-199412000-00002. PMID 7712044
- [Background] Austin MA. Small, dense low-density lipoprotein as a risk factor for coronary heart disease. Int J Clin Lab Res. 1994;24(4):187-92. doi: 10.1007/BF02592460. PMID 7894041
- [Background] Austin MA. Genetic and environmental influences on LDL subclass phenotypes. Clin Genet. 1994 Jul;46(1 Spec No):64-70. doi: 10.1111/j.1399-0004.1994.tb04204.x. PMID 7988081
- [Background] Austin MA, Hokanson JE. Epidemiology of triglycerides, small dense low-density lipoprotein, and lipoprotein(a) as risk factors for coronary heart disease. Med Clin North Am. 1994 Jan;78(1):99-115. doi: 10.1016/s0025-7125(16)30178-x. PMID 8283937
- [Background] Austin MA, Jarvik GP, Hokanson JE, Edwards K. Complex segregation analysis of LDL peak particle diameter. Genet Epidemiol. 1993;10(6):599-604. doi: 10.1002/gepi.1370100645. PMID 8314067